CLINICAL TRIAL: NCT04520581
Title: The Use of "O" Shaped- Endotracheal Tube During Intubation for General Anesthesia: Prospective Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yu-Kyung Bae, clinical professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: B-2003-603-304
Record Dates: First submitted 2020-08-13; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Endotracheal Intubation
MeSH Terms: interventions — O-antigen, Acinetobacter strain 90

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Use in the shape of an endotracheal tube.
- Group "O" (Experimental): Just before the induction of medicine is injected, the assistant makes endotracheal tube into "O" shape.
  Interventions: Other: group "O"

INTERVENTIONS:
Other: group "O" — Endotracheal tube was made "O" shape by assistants.
  Arms: Group "O"

SUMMARY:
This study is prospective randomized trial study. "O" type tracheal intubation tube is anatomically consistent and will able to increase the success rate of first intubation without any other external help.

DETAILED DESCRIPTION:
This study is divided into two groups. : control vs. "O" shape endotracheal tube.

The investigator was studied 238 consecutive the American Society of Anesthesiologists' physical grades I and II adult patients scheduled to undergo general anesthesia requiring tracheal intubation for elective surgery. Exclusion criteria included a gross anatomical abnormality, before surgery of the head, neck and cervical spine, previously difficult tracheal intubation, loose teeth, or those requiring a rapid sequence or awake intubation, moderate or severe obstructive/restrictive pulmonary disease accompanied by pulmonary function tests. Anesthesia was induced with remifentanyl 3ng/kg, propopol 1-2 mg/kg or TIVA 2% fresopol 4ug/dL, remifentanyl 3ng/dL and rocuronium 0.8 mg/kg to facilitate tracheal intubation. Laryngoscopy was performed after the loss of the fourth twitch in the train-of-four in response to ulnar nerve stimulation. All laryngoscopies using a #4 Macintosh blade were performed with the patient placed in the sniffing position. Tracheal intubation was performed without assistance (ex. External laryngeal manipulation, Used stylet). A single experienced anesthesiologist, blinded to each group, performed all of the direct laryngoscopies and classified the laryngoscopic view according to the modified Cormack and Lehane grade, measured number of attempts, intubation time and blood pressure and heart rate before/ after intubation.

ELIGIBILITY:
Inclusion Criteria:

* Consented to participate in the study
* Aged 19 years or older
* The American Society of Anesthesiologists' physical grades I and II
* Undergo elective surgery under general anesthesia

Exclusion Criteria:

* Do not agree to participate in research
* Previously difficult tracheal intubation
* Rapid induction of anesthesia
* Previous c-spine disc or had surgery
* Teeth are severely shaken or poor
* Moderate or severe obstructive/restrictive pulmonary disease accompanied by pulmonary function tests

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
First intubation success rate for each between two group | Immediately after intubation
  First laryngoscope tries was success using detection of end tidal CO2

SECONDARY OUTCOMES:
First intubation time | within 60 seconds
  After intubation, appearing end tidal CO2 at monitoring
Number of attempts | From the first tracheal intubation failure to the next successful tracheal intubation
  Number of intubation try
Measured vital sign | immediately before intubation and within 5 minites after intubation
  Blood pressure in mmHg and heart rate in bpm were recorded immediately before and after intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kyung Bae, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeongggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No